CLINICAL TRIAL: NCT04531072
Title: Effect of Atazanavir-ritonavir on the Pharmacokinetics and Toxicity of Lumefantrine in People Living With HIV Attending Lagos University Teaching Hospital
Brief Title: Effect of Atazanavir-ritonavir on the Pharmacokinetics and Toxicity of Lumefantrine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fogarty International Center of the National Institute of Health (NIH)
Collaborators: NIH Office of AIDS Research (OAR) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Sikiru Olatunji Usman, Principal Investigator, Fogarty International Center of the National Institute of Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D43TW010134 (NIH)
Record Dates: First submitted 2020-08-16; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Drug Interaction
Keywords: Drug interaction, artemether-lumefantrine, atazanavir-ritonavir, LUTH
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination; atazanavir, ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Two arm study namely: ATVr arm and AL (Control) arm each consisting of 10 participants in a parallel study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ATVr-arm (Experimental): 10 participants living with HIV and having uncomplicated Falciparum malaria were administered: Atazanavir-ritonavir (300/100 mg) one tablet once daily continuously + tenofovir-lamivudine (300/300 mg) one tablet once daily continuously and artemether-lumefantrine (80/480 mg) one tablet twice daily for three days at 0, 8, 24, 36, 48 and 60 hour.
  Interventions: Drug: Artemether-lumefantrine; Drug: Atazanavir-ritonavir 300/100 mg
- AL-arm (Control) (Active Comparator): 10 participants who were HIV negative but having uncomplicated Falciparum malaria were administered: Artemether-lumefantrine 80/480 mg, one tablet twice daily for three days at 0, 8, 24, 36, 48 and 60 hour.
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Safety and efficacy evaluation during concurrent use of artemether-lumefantrine and atazanavir-ritonavir based antiretroviral therapy
  Other Names: Coartem 80/480, P01BF01
Drug: Atazanavir-ritonavir 300/100 mg — Safety and efficacy evaluation during concurrent use of artemether-lumefantrine and atazanavir-ritonavir based antiretroviral therapy
  Other Names: Anzavir-R, J05AR23
  Arms: ATVr-arm

SUMMARY:
A case control pharmacokinetic study evaluating the effects of atazanavir-ritonavir on the pharmacokinetics and toxicity of lumefantrine in people living with HIV attending APIN clinic of the Lagos University Teaching Hospital

DETAILED DESCRIPTION:
Atazanavir-ritonavir (ATVr) based antiretroviral therapy and artemether-lumefantrine (AL) are commonly used drugs for the treatment of Human Immune Deficiency Virus (HIV) infection and malaria respectively in Nigeria. However, both drugs interact with Cytochrome P 3A4 (CYP 3A4) isoenzymes which may spawn clinically significant pharmacokinetic interactions.

The study was aimed at evaluating the effects of atazanavir-ritonavir on the pharmacokinetics and toxicity of lumefantrine.

In a case control pharmacokinetic study, twenty participants who tested positive for Plasmodium falciparum malaria were recruited and divided into two groups (ATVr-arm, n=10; and Control-arm, n= 10). All the participants were administered with 6 doses of AL 80-480 mg (Coartem). Thereafter, blood samples were collected from them at different time intervals over seven days. The lumefantrine concentration in each sample was determined with high-performance liquid chromatography (HPLC) and entered into WinNonlin® software to determine the pharmacokinetic parameters of lumefantrine which were compared between the test and control groups. Toxicity was evaluated with adverse events monitoring, electrocardiography, haematological and blood chemistry tests at pre and post doses of artemether-lumefantrine.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-gravid female ≥18 years of age,
* Informed written consent,
* Malaria parasitaemia
* Axillary temperature ≥37.5°C or history of fever within 24 hours before visiting the clinic and with, at least, any of the following signs and symptoms of uncomplicated malaria: chills, sweats, headaches, muscle aches, nausea, vomiting, diarrhoea, body weakness, poor appetite and pallor.
* Hemoglobin (Hb) ≥8 g/dl
* Body weight ≥35 kg
* HIV positive (ATVr arm), HIV negative (AL/control arm)

Exclusion Criteria:

* Severe anaemia' (Haemoglobin levels < 8g/dl)
* Smokers/alcoholics and users of substances which inhibit or induce CYP3A4 iso enzymes
* Withdrawal of consent
* Known allergy to any of the study drugs
* Development of complications or severe adverse effects
* Smokers/alcoholics and users of caffeine, drugs which induce or inhibit CYP3A4 and CYP2B6
* Evidence of chronic illnesses such as diabetes, hypertension, psychiatric illnesses
* Subject taking any drugs or having any condition known to prolong QT-intervals
* Signs of severe malaria
* Use of anti-tubercular drugs for at least three months prior to enrolment
* Being on anti-malarial drugs within four weeks prior to enrolment
* Pregnant or nursing mother.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Drug exposure (Area under the curve) of lumefantrine | 2 weeks
  Change in drug exposure (AUC) of lumefantrine may indicate interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction
Maximum plasma concentration (Cmax) of lumefantrine | 2 weeks
  Change in maximum plasma concentration (Cmax) of lumefantrine may indicate interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction
Day 7 lumefantrine concentration | 2 weeks
  This the plasma concentration of lumefantrine at the seventh day of commencement of the first dose. Efficacy is indicated when it is 280 ng/mL and above.
QTc-interval | One week
  Change in mean or median QTc-interval above therapeutic range at post-dose of artemether-lumefantrine indicates cardio-toxicity caused by interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction.
Haemoglobin level | One week
  Change in mean or median hemoglobin level above therapeutic range at post-dose of artemether-lumefantrine indicates haemotoxicity caused by interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction.
Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels | One week
  Change in mean or median ALT and AST levels above therapeutic range at post-dose of artemether-lumefantrine indicates liver toxicity caused by interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction.
Creatinine level | One week
  Change in mean or median creatinine level above therapeutic range at post-dose of artemether-lumefantrine indicates renal toxicity caused by interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction.
Adverse events | Two weeks
  Change in frequency of adverse events post-dose of artemether-lumefantrine indicates toxicity caused by interaction between atazanavir-ritonavir and lumefantrine via Cytochrome P3A4 induction.

CONTACTS AND LOCATIONS:
Overall Officials: Sikiru Usman, Ph.D., Principal Investigator — University of Lagos; Ibrahim Oreagba, Ph.D., Study Director — University of Lagos
Locations (1):
- Apin (Aids Prevention Initiatives in Nigeria) clinic, Lagos University Teaching Hospital, Surulere, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No
IPD would not be made available to other researchers

REFERENCES:
- [Derived] Usman SO, Oreagba IA, Kadri MR, Adewumi OO, Akinyede A, Agbaje EO, Abideen G, Busari AA, Hassan OO, Akinleye MO, Akanmu AS. Evaluation of the effects of atazanavir-ritonavir on the pharmacokinetics of lumefantrine in patients living with HIV in Lagos University Teaching Hospital, South-Western Nigeria. Eur J Clin Pharmacol. 2021 Sep;77(9):1341-1348. doi: 10.1007/s00228-021-03116-x. Epub 2021 Mar 23. PMID 33755736